CLINICAL TRIAL: NCT03375866
Title: Effects of Mixed Nut Consumption on Satiety and Weight Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2515098
Record Dates: First submitted 2017-12-11; First posted 2017-12-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Satiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pretzels (Active Comparator)
  Interventions: Other: Pretzels
- Mixed nuts (Experimental)
  Interventions: Other: Mixed nuts

INTERVENTIONS:
Other: Pretzels — Subjects consume 240 kcal of pretzels daily for 16 weeks.
  Arms: Pretzels
Other: Mixed nuts — Subjects consume 240 kcal of mixed nuts daily for 16 weeks.
  Arms: Mixed nuts

SUMMARY:
The first goal of the proposed study is to determine acute and long-term effects of mixed nuts (almonds, hazelnuts, pecans, pistachios, walnuts, and peanuts) on metabolic parameters and weight management. While numerous studies have shown the beneficial effects of nuts on promoting negative energy balance and weight loss, mechanistic studies exploring how the inclusion of nuts in the diet promotes a negative energy balance and weight loss have not been conducted. The second goal is to determine the mechanisms by which mixed nut consumption regulates of food intake and body weight.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old
* BMI 27-40

Exclusion Criteria:

* Smoker
* Pregnant woman
* Required dietary supplement use
* Required medication of metabolic disorders
* Allergy to nuts or gluten

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change of Satiety | 0, 20, 40, 60, 90 and 120 minutes post snack consumption
  Hunger feeling (appetite) will be examined using visual analog scale (0-10): 0 least and 10 greatest
Change of glucose level | Baseline, 40 minutes post snack consumption, and 8 weeks and 16 weeks post daily consumption
  Glucose level will be examined using glucose analysis
Change of insulin level | Baseline, 40 minutes post snack consumption, and 8 weeks and 16 weeks post daily consumption
  Insulin level will be examined using an ELISA biochemical method
Change of cholesterol levels | 8 weeks and 16 weeks post daily consumption
  Cholesterol levels will be examined using a biochemical method
Change of Lp(a) | 8 weeks and 16 weeks post daily consumption
  Lp(a) levels will be examined using an ELISA biochemical method

SECONDARY OUTCOMES:
Change of microbiome | 8 weeks and 16 weeks post daily consumption
  Diversity of microbiome will be analyzed in fecal samples

CONTACTS AND LOCATIONS:
Locations (1):
- School of Exercise and Nutritional Sciences, SDSU, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nora CL, Zhang L, Castro RJ, Marx A, Carman HB, Lum T, Tsimikas S, Hong MY. Effects of mixed nut consumption on LDL cholesterol, lipoprotein(a), and other cardiometabolic risk factors in overweight and obese adults. Nutr Metab Cardiovasc Dis. 2023 Aug;33(8):1529-1538. doi: 10.1016/j.numecd.2023.05.013. Epub 2023 May 15. PMID 37263914
- [Derived] Rosas M Jr, Liu C, Hong MY. Effects of Mixed Nut Consumption on Blood Glucose, Insulin, Satiety, and the Microbiome in a Healthy Population: A Pilot Study. J Med Food. 2023 May;26(5):342-351. doi: 10.1089/jmf.2022.0121. Epub 2023 Apr 20. PMID 37083461